CLINICAL TRIAL: NCT01933373
Title: A Prospective Randomized Trial Comparing Two Reconstructive Operation Techniques After Myotomy of Achalasia. Comparing Toupet Versus DOR.
Brief Title: A Prospective Study Comparing Two Reconstructive Operation Techniques After Myotomy of Achalasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Ersta Hospital, Sweden (Other)
Responsible Party: Principal Investigator, Lars Lundell, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/595-32
Record Dates: First submitted 2013-06-19; First posted 2013-09-02 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Achalasia
Keywords: Randomized; Toupet; Dor; Achalasia
MeSH Terms: conditions — Esophageal Achalasia | interventions — Myotomy; Receptors, Opioid, delta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toupet (Active Comparator): Laparoscopic Myotomy + Toupet 180 degree partial posterior fundoplication.
  Interventions: Procedure: Toupet
- Dor (Experimental): Laparoscopic Myotomy + Dor anterior partial fundoplication. 90 degree partial fundoplication being the standard of care.
  Interventions: Procedure: Dor

INTERVENTIONS:
Procedure: Toupet — Laparoscopic posterior partial fundoplication plus myotomy.
  Other Names: Laparascopic posterior partial fundoplication plus myotomy.
  Arms: Toupet
Procedure: Dor — Anterior partial fundoplication plus myotomy.
  Other Names: Anterior partial fundoplication plus myotomy.
  Arms: Dor

SUMMARY:
Achalasia is a rare motor disorder of the gastroesophageal junction which is associated with an increased pressure of the esophageal sphincter. This leads to impairment to swallow and heartburn. Esophageal myotomy, which is a surgical longitudinal incision of the esophageal muscle layer extending over to the gastroesophageal junction is the treatment of choice for achalasia. In order to prevent reflux of stomach content into the esophagus this has to be combined with an antireflux procedure where the upper part of the stomach (fundus) is wrapped around the esophagus (fundoplication). This procedure can be performed with the wrapped fundus either in front of the esophagus (Dor procedure) or behind (Toupet). The latter introduces an angulation of the esophagus, which possibly may lead to an impairment of swallowing ability and passage of food to the stomach. On the other hand, the Toupet procedure may give a better control of reflux. The primary endpoint of the study is symptoms of impaired swallowing 1 year after treatment. Secondary outcomes include reflux (pH measurements in the esophagus), radiological imaging of swallowing and quality of life.

DETAILED DESCRIPTION:
By the end of 2012 40 patients have been enrolled and passed the one year follow up.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Typical achalasia according to manometry
* Eckhardt score >3
* Informed consent

Exclusion Criteria:

* Severe comorbidity precluding surgery
* Pseudo achalasia
* Inability to participate in follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-05; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Dysphagia symptoms according to Eckhardt | up to five years follow up

SECONDARY OUTCOMES:
Ambulatory esophageal PH | One and five years follow up
Health-related quality of life according to Velanovich | One and five years follow up
Timed barium esophagogram at 1, 2 and 5 minutes | One and five years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Lars R Lundell, Professor, Principal Investigator — Gastrocentrum Karolinska University Hospital, Stockholm Sweden
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Kumagai K, Kjellin A, Tsai JA, Thorell A, Granqvist S, Lundell L, Hakanson B. Toupet versus Dor as a procedure to prevent reflux after cardiomyotomy for achalasia: results of a randomised clinical trial. Int J Surg. 2014;12(7):673-80. doi: 10.1016/j.ijsu.2014.05.077. Epub 2014 Jun 2. PMID 24892729